CLINICAL TRIAL: NCT06729970
Title: A Phase 1, 6-part, Open-label, Fixed-sequence Study to Evaluate the Effects of Lithium, Valproic Acid, and Lamotrigine on the Single-dose Pharmacokinetics of KarXT and Effects of KarXT on the Single-dose Pharmacokinetics of Lithium, Valproic Acid, and Lamotrigine in Healthy Participants
Brief Title: A Study to Evaluate the Effects of Lithium, Valproic Acid, and Lamotrigine on the Pharmacokinetics of KarXT and Effects of KarXT on the Pharmacokinetics of Lithium, Valproic Acid, and Lamotrigine in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Karuna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CN012-0035
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers
Keywords: KarXT; Lithium; Valproic acid; Drug-Drug Interaction study; Healthy Volunteers; BMS-986510; Pharmacokinetics; Lamotrigine
MeSH Terms: interventions — xanomeline; trospium chloride; Lithium; Valproic Acid; Lamotrigine

STUDY DESIGN:
Intervention Model Description: Parallel A & B cohorts, then Parallel C & D cohorts and then parallel E&F cohorts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A (Experimental)
  Interventions: Drug: Xanomeline/Trospium Chloride; Drug: Lithium
- Part B (Experimental)
  Interventions: Drug: Xanomeline/Trospium Chloride; Drug: Valproic Acid
- Part C (Experimental)
  Interventions: Drug: Xanomeline/Trospium Chloride; Drug: Lithium
- Part D (Experimental)
  Interventions: Drug: Xanomeline/Trospium Chloride; Drug: Valproic Acid
- Part E (Experimental)
  Interventions: Drug: Xanomeline/Trospium Chloride; Drug: Lamotrigine
- Part F (Experimental)
  Interventions: Drug: Xanomeline/Trospium Chloride; Drug: Lamotrigine

INTERVENTIONS:
Drug: Xanomeline/Trospium Chloride — Specified dose on specified days
  Other Names: BMS-986510; KarXT
Drug: Lithium — Specified dose on specified days
  Arms: Part A; Part C
Drug: Valproic Acid — Specified dose on specified days
  Arms: Part B; Part D
Drug: Lamotrigine — Specified dose on specified days
  Arms: Part E; Part F

SUMMARY:
The purpose of this study is to evaluate the effects of lithium, valproic acid, and lamotrigine on the single-dose pharmacokinetics (PK) of KarXT and the effect of KarXT on the single-dose PK of lithium, valproic acid, and lamotrigine in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female [individual not of childbearing potential (INOCBP)] participants as determined by no clinically significant deviation from normal in medical history, physical examination, 12-lead ECG, vital signs, and clinical laboratory determinations.
* BMI of 18.0 to 32.0 kg/m2, inclusive.

Exclusion Criteria:

* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, GI, endocrine, immunologic, dermatologic, neurologic, or oncologic disease or any other condition that, in the opinion of the investigator, would jeopardize the safety of the participant or the validity of the study results. Note: Any grade of hepatic impairment (Child-Pugh Grade A or higher) is excluded.
* Parts B and D only: History of pancreatitis.
* Any significant acute or chronic medical illness, in the opinion of the investigator.
* History or high risk of urinary retention, gastric retention, or narrow-angle glaucoma or known history of prostate hypertrophy or nocturia.
* Parts E & F only: history of skin rash and mucus ulcerations of no obvious cause and Gilbert's syndrome
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-12-26 (Actual); Primary Completion 2026-01-18 (Estimated); Study Completion 2026-01-18 (Estimated)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to day 54
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC(0-T)) | Up to day 54
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) | Up to day 54

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 28 days post discontinuation of dosing
Number of participants with serious adverse events (SAEs) | Up to 28 days post discontinuation of dosing
Number of participants with physical examination abnormalities | Up to 2 days post discontinuation of dosing
Number of participants with vital sign abnormalities | Up to 2 days post discontinuation of dosing
Number of participants with 12-lead electrocardiogram (ECG) abnormalities | Up to 2 days post discontinuation of dosing
Number of participants with clinical laboratory abnormalities | Up to 2 days post discontinuation of dosing
Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to 2 days post discontinuation of dosing
Number of participants with AEs of Special Interest (AESIs) | Up to 28 days post discontinuation of dosing

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- CenExel Collaborative Neuroscience Research, LLC - Los Alamitos, Los Alamitos, California, United States

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06729970.html